CLINICAL TRIAL: NCT03652636
Title: Evaluation of the Efficacy of Contrast Enhanced Ultrasound Compared to MRI for Differentiation of Hepatic Lesions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Jordan K. Swensson, Assistant Professor of Clinical Radiology and Imaging Sciences, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RADY-SWENSSON
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Hepatic Disease
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- One: Patient population with hepatic lesion(s) (Other): Patient scheduled to get MRI will also be asked to receive an ultrasound of the liver
  Interventions: Drug: Sulfur Hexafluoride Microspheres

INTERVENTIONS:
Drug: Sulfur Hexafluoride Microspheres — 2.5 mL intravenous injection given at the time of ultrasound, with second 2.5 mL intravenous injection given during ultrasound as needed to improve visualization
  Other Names: Lumason

SUMMARY:
In patients with hepatic lesions, to evaluate the efficacy of contrast enhanced ultrasound compared to MRI in differentiating focal nodular hyperplasia and hepatic adenoma.

DETAILED DESCRIPTION:
Hepatic imaging plays an important role in identifying and differentiating both benign and malignant neoplasms of the liver. One of the clinical and radiologic dilemmas facing hepatic medicine is the accurate differentiation of focal nodular hyperplasia (FNH) and hepatic adenoma (HA). This is a question of some import, as there are significant prognosis and treatment differences between these entities, as well as overlap in the patient populations in whom they occur.

FNH is the second most common benign neoplasm of the liver, with a strong female predilection. These lesions are usually asymptomatic and incidentally discovered, and carry only a small risk of complication such as bleeding. There is no malignant potential. Hepatic adenomas (HAs) are more rare benign neoplasms that also have a female predilection. However, these lesions are more likely to be symptomatic, and carry a higher bleeding risk especially as they grow over 4 cm. In addition, they harbor a small risk of malignant transformation to hepatocellular carcinoma (HCC). Of note, patients may present with both types of lesion concurrently.

Currently, MRI with hepatobiliary contrast agents is the standard for differentiation of these lesions. These agents (such as gadoxetate disodium, or Eovist) are actively transported into hepatocytes, which are present in FNH and only in very rare cases with HA. Previous research (such as from Grazioli et al.) has shown that hepatobiliary agents can differentiate these lesions with excellent accuracy. However, there is still overlap between these lesions on imaging, and for certain patients MRI may be difficult or impossible.

FDA approval of contrast enhanced ultrasound (CEUS) agents in 2016 has opened a new avenue for abdominal imaging. CEUS utilizes gas containing lipid microbubbles to provide pure intravascular contrast, allowing for evaluation of vascular and solid organ perfusion. It has an excellent safety profile and is not excreted by the kidneys, allowing for use in patients with acute and chronic renal disease. It has been used for some time outside of the US for liver lesion evaluation, and the enhancement patterns of both FNH and HA have been described in the literature by Kim et al. as having different appearances. CEUS can be especially useful for focal liver lesion imaging for patients who cannot or will not undergo MRI, and it has the advantages of flexibility, increased temporal resolution, and decreased cost. This study aims to compare the utility of CEUS for differentiating FNH and HA with the current standard of hepatobiliary contrast MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females
2. Age 18 years or greater
3. Scheduled to undergo abdominal MRI with contrast at a performance site for evaluation of a hepatic lesion(s).

Exclusion criteria:

1. History of cardiac shunting
2. History of acute cardiac ischemia
3. History of hypersensitivity reaction to Lumason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan K Swennson, MD, Principal Investigator — Indiana University
Locations (1):
- IU University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swensson J, McCrate M, Halappa VG, Stethen T, Akisik F. Contrast-Enhanced Ultrasound Compared With Hepatobiliary Agent MRI for Differentiation of Focal Nodular Hyperplasia and Hepatic Adenoma: A Prospective Trial. Ultrasound Q. 2024 Nov 22;40(4):e00696. doi: 10.1097/RUQ.0000000000000696. eCollection 2024 Dec 1. PMID 39589314

RESULTS

PARTICIPANT FLOW:
Groups:
- =Patient Population With Liver Lesion(s): Patients with hepatic lesion(s) scheduled to get MRI will also be asked to receive an ultrasound of the liver. Sulfur Hexafluoride Microspheres (2.5 mL) intravenous injection will be given at the time of ultrasound, with second 2.5 mL intravenous injection given during ultrasound as needed to improve visualization.
Period: Overall Study
Arm/Group | =Patient Population With Liver Lesion(s)
Started | 47
Completed | 40
Not Completed | 7
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Groups:
- =Patient Population With Liver Lesion(s): 40 patients with liver lesion(s) identified in MRI
Arm/Group | =Patient Population With Liver Lesion(s)
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of CEUS at Differentiating Focal Nodular Hyperplasia (FNH) From Hepatocellular Adenoma (HCA)
Description: To compare the ability of contrast enhanced ultrasound to differentiate between hepatic adenoma and FNH compared with the current standard of contrast enhanced MRI.
Time Frame: One day
Population: 59 liver lesions were evaluated with a one time contrast enhanced ultrasound. Two blinded radiologists then evaluated the CEUS images and gave a diagnosis of FNH or HCA
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Liver lesions
Groups:
- Reader 1 - CEUS Sensitivity / Specificity Differentiating FNH & HCA; Reader 2 - CEUS Sensitivity / Specificity Differentiating FNH & HCA: Patients with hepatic lesion(s) scheduled to get MRI will also be asked to receive an ultrasound of the liver. Sulfur Hexafluoride Microspheres (2.5 mL) intravenous injection will be given at the time of ultrasound, with second 2.5 mL intravenous injection given during ultrasound as needed to improve visualization
Arm/Group | Reader 1 - CEUS Sensitivity / Specificity Differentiating FNH & HCA | Reader 2 - CEUS Sensitivity / Specificity Differentiating FNH & HCA
Number analyzed (Participants) | 40 | 40
Number analyzed (Liver lesions) | 59 | 59
percentage of lesions
  Sensitivity (true positive rate) | 66.7 | 64.0
  Specificity (true negative rate) | 71.9 | 90.6
  Accuracy (is the ultrasound assessment of the lesion correct) | 69.5 | 78.0

2. Secondary Outcome: AUC of Differentiating FNH From HCA (AUC Represents the Probability That the Model, if Given a Randomly Chosen Correct and Incorrect CEUS Diagnosis of a Lesion, Will Rank the Correct Higher Than the Incorrect)
Description: To compare the ability of contrast enhanced ultrasound to differentiate FNH from HCA
Time Frame: One day
Population: as for outcome 1
Measure: Number; unit: Probability of correct evaluation
Units Other Than Participants: liver lesions
Arm/Group | Reader 1 - CEUS Sensitivity / Specificity Differentiating FNH & HCA | Reader 2 - CEUS Sensitivity / Specificity Differentiating FNH & HCA
Number analyzed (Participants) | 40 | 40
Number analyzed (liver lesions) | 59 | 59
Probability of correct evaluation | 0.693 | 0.768

ADVERSE EVENTS:
Time Frame: One day
Description: Reporting uses standard definitions
Arm/Group | =Patient Population With Liver Lesion(s)
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT03652636/Prot_002.pdf
  • Statistical Analysis Plan (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT03652636/SAP_003.pdf
  • Informed Consent Form (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT03652636/ICF_004.pdf